CLINICAL TRIAL: NCT01431391
Title: A Randomized, Open-Label, Phase 2 Trial Examining the Sequencing of Sipuleucel-T and Androgen Deprivation Therapy in Men With Non-metastatic Prostate Cancer and a Rising Serum Prostate Specific Antigen After Primary Therapy
Brief Title: Sequencing of Sipuleucel-T and ADT in Men With Non-metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P10-2
Record Dates: First submitted 2011-08-05; First posted 2011-09-09 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Prostatic Neoplasm; Prostate Cancer; Prostatic Adenocarcinoma
Keywords: Immune therapy; Cancer vaccine; Therapeutic vaccine; Therapeutic cancer vaccine; Vaccine; Dendritic cells; PSA; Androgen deprivation therapy; Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms; Prostatic Diseases; Androgens; Hormones; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial; Immunology; Hormone therapy; Immunotherapy; Luteinizing hormone-releasing hormone (LHRH)
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms; Prostatic Diseases; Adenocarcinoma; Carcinoma; Neoplasms, Glandular and Epithelial | interventions — sipuleucel-T; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Sipuleucel-T followed by ADT (Experimental): Arm 1: Subjects received one infusion of sipuleucel-T every two weeks for a total of three infusions. Two weeks after the third sipuleucel-T infusion, subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg). An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT.
  Interventions: Biological: sipuleucel-T; Drug: leuprolide acetate
- Arm 2: ADT followed by sipuleucel-T (Experimental): Arm 2: Subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg) 12 weeks before infusion 1 of sipuleucel-T. An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT. Twelve weeks after the initial leuprolide 45 mg depot injection, subjects began one infusion of sipuleucel-T every two weeks for a total of three infusions.
  Interventions: Biological: sipuleucel-T; Drug: leuprolide acetate

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF).
  Other Names: PROVENGE®; APC8015
Drug: leuprolide acetate — 45.0 mg depot injection, 2 doses 6 months apart
  Other Names: Eligard®

SUMMARY:
The main purpose of this study was to determine whether ADT started before or after sipuleucel-T led to a better immune system response. This study also evaluated the safety of sipuleucel-T and ADT treatment, immune system responses over time, the characteristics of sipuleucel-T, and changes in prostate specific antigen (PSA) values over time.

DETAILED DESCRIPTION:
Multicenter, randomized, open-label study, with subjects allocated (1:1) to 1 of 2 study arms, using a stratified randomization based on:

• Prostate-specific antigen doubling time (PSADT): ≤ 3 months or > 3 months and ≤ 12 months. • Primary therapy: radical prostatectomy (RP) or radiation, including brachytherapy, (XRT) or RP + XRT.

Arm 1: Subjects received one infusion of sipuleucel-T every two weeks for a total of three infusions. Two weeks after the third sipuleucel-T infusion, subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg). An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT.

Arm 2: Subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg) 12 weeks before infusion 1 of sipuleucel-T. An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT. Twelve weeks after the initial leuprolide 45 mg depot injection, subjects began one infusion of sipuleucel-T every two weeks for a total of three infusions.

Cellular and humoral immune responses were assessed for Arm 2 subjects at 12, 8, and 4 weeks pre infusion 1, and in all subjects (both arms) at pre-leukapheresis 1, 2, and 3, and post-infusion 1, 2 and 3, and at the following time points after the third infusion: Weeks 2, 6, and 12 and Months 6, 9, 12, 15, 18, 21, and 24.

Safety assessments included adverse event (AE) monitoring, laboratory tests (complete blood count (CBC) and serum chemistry), vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, as well PSA and testosterone monitoring. The study was complete at the 27-Month visit for Arm 1 and the 24-Month visit for Arm 2.

ELIGIBILITY:
Inclusion Criteria:

* Hormone-sensitive prostate cancer
* Non-metastatic disease, as evidenced by negative bone scan or computed tomography of the abdomen and pelvis
* ECOG performance status ≤ 1
* Histologically documented prostate cancer
* Prior primary therapy for prostate cancer
* Rising PSA with a PSADT of ≤ 12 months
* Testosterone ≥ 200 ng/dL ≤ 28 days of registration
* Adequate hematologic, renal, and liver function
* Must live in a permanent residence within a comfortable driving distance (round-trip within one day) to the clinical research site

Exclusion Criteria:

* Requires systemic ongoing immunosuppressive therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sipuleucel-T or GM-CSF
* Prior sipuleucel-T therapy
* Prior ADT therapy ≤ 6 months prior to registration or ≥ 6 months duration in total
* If subject has a history of any other stage III/IV malignancy, the subject must be disease free and off any malignancy-related treatment for at least 10 years. If the subject has a history of any stage I-II malignancy, the subject must be disease free and off any malignancy-related treatment for at least 5 years.
* Prior experimental immunotherapy or on an experimental clinical trial within 1 year
* Received denosumab or XRT ≤ 6 months prior to registration
* Received chemotherapy or GM-CSF ≤ 90 days prior to registration
* Received any of the following medications or interventions ≤ 28 days prior to registration

  * major surgery requiring general anesthesia
  * systemic immunosuppressive therapy
  * other prescription treatment for prostate cancer
* Active infection within 1 week of registration
* Likely to receive XRT or surgery for prostate cancer during the study period
* Any medical intervention, any other condition, or any circumstances that could compromise the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (14):
- United States (14):
  - Urology Center of Alabama, Homewood, Alabama
  - University of California San Diego / Moores Cancer Center, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - The Urology Center of Colorado, Denver, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NYOH Albany Cancer Center at Patroon Creek, Albany, New York
  - Community Care Physicians, PC, Albany, New York
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology San Antonio Research, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1:Sipuleucel-T Followed by ADT: Subjects received one infusion of sipuleucel-T every two weeks for a total of three infusions. Two weeks after the third sipuleucel-T infusion, subjects started androgen deprivation therapy (ADT) with 45 mg leuprolide acetate depot injection (Eligard® 45 mg). An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT.
- Arm 2: ADT Followed by Sipuleucel-T: Subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg) 12 weeks before infusion 1 of sipuleucel-T. An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT. Twelve weeks after the initial leuprolide 45 mg depot injection, subjects began one infusion of sipuleucel-T every two weeks for a total of three infusions.
Period: Overall Study
Arm/Group | Arm 1:Sipuleucel-T Followed by ADT | Arm 2: ADT Followed by Sipuleucel-T
Started | 34 | 34
Received ≥1 Leaukapheresis | 34 | 34
Completed | 26 | 30
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Sipuleucel-T Followed by ADT: Subjects received one infusion of sipuleucel-T every two weeks for a total of three infusions. Two weeks after the third sipuleucel-T infusion, subjects started ADT with 45 mg leuprolide acetate depot injection (Eligard® 45 mg). An additional leuprolide acetate injection was administered at 6 months after the first injection for a total of 2 injections and 12 months of ADT.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Sipuleucel-T Followed by ADT | Arm 2: ADT Followed by Sipuleucel-T | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (1.4) | 66.2 (1.1) | 65.8 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 34 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions. | 33 | 34 | 67
    ECOG 1= Restricted Strenuous Activity | 1 | 0 | 1
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤ 6 | 3 | 4 | 7
    Gleason Score = 7 | 23 | 21 | 44
    Gleason Score ≥ 8 | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Immune Response at Month 24 as Evaluated by IFN-γ ELISPOT Specific for PA2024
Description: Immune response at month 24 as evaluated by IFN-γ ELISPOT specific for PA2024 following sipuleucel-T/ADT treatment regimens to determine if order of administration impacted immune response.
Time Frame: PA2024 ELISPOT counts at Month 24
Population: The immune response population was defined as all randomized subjects who received 3 infusions of sipuleucel-T.
Measure: Mean (Standard Error); unit: IFN-γ ELISPOT (per 300,000 PBMC)
Arm/Group | Arm 1: Sipuleucel-T Followed by ADT | Arm 2: ADT Followed by Sipuleucel-T
Number analyzed (Participants) | 19 | 26
IFN-γ ELISPOT (per 300,000 PBMC) | 81.0 (28.0) | 61.1 (23.7)

2. Secondary Outcome: Percentage of Participants With Immune Response As Evaluated by IFN-γ ELISPOT Specific for PA2024
Description: A participant was considered to have an immune response it the post-baseline PA2024-specific IFN-g ELISPOT count was >18
Time Frame: Month 24
Population: The immune response population was defined as all randomized subjects who received 3 infusions of sipuleucel-T.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1:Sipuleucel-T Followed by ADT | Arm 2: ADT Followed by Sipuleucel-T
Number analyzed (Participants) | 33 | 34
percentage of participants | 88 | 85

ADVERSE EVENTS:
Time Frame: All non-serious adverse events (AE)s and serious adverse events (SAE)s, were collected at all visits through Month-6 or at early withdrawal.
Description: Following Month-6 only possible or probable treatment-related AEs and cerebrovascular events (CVE)s were recorded: Months 9, 12, 15, 18, 21, 24 (and 27 in Arm 1). Adverse events are reported in the safety population defined as subjects who received at least one leukapheresis.
Arm/Group | Arm 1: Sipuleucel-T Followed by ADT | Arm 2: ADT Followed by Sipuleucel-T
Serious Adverse Events (participants affected / at risk) | 1/34 | 5/34
Other Adverse Events (participants affected / at risk) | 33/34 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Sipuleucel-T Followed by ADT (N=34) | Arm 2: ADT Followed by Sipuleucel-T (N=34)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Device-related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Sipuleucel-T Followed by ADT (N=34) | Arm 2: ADT Followed by Sipuleucel-T (N=34)
Hot flush (Vascular disorders) | 19 (20) | 23 (23)
Fatigue (General disorders) | 13 (19) | 21 (26)
Headache (Nervous system disorders) | 9 (10) | 7 (7)
Chills (General disorders) | 9 (19) | 6 (8)
Citrate toxicity (Injury, poisoning and procedural complications) | 6 (12) | 6 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (4)
Paraesthesia oral (Gastrointestinal disorders) | 5 (9) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Contusion (Injury, poisoning and procedural complications) | 5 (6) | 3 (4)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Weight increased (Investigations) | 4 (4) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 6 (7)
Oedema peripheral (General disorders) | 3 (3) | 4 (4)
Haematoma (Vascular disorders) | 3 (4) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 3 (5) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (6) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 1 (1)
Influenza-like illness (General disorders) | 0 (0) | 3 (4)
Infusion-related reaction (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Injection-site extravasation (General disorders) | 1 (1) | 2 (2)
Injection-site haematoma (General disorders) | 1 (1) | 2 (3)
Micturation urgency (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Loss of libido (Psychiatric disorders) | 0 (0) | 2 (2)
Libido decreased (Psychiatric disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 2 (4)
Urinary retention (Renal and urinary disorders) | 2 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 5 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (7)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Paraesthesia (Nervous system disorders) | 5 (5) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.